CLINICAL TRIAL: NCT06032130
Title: "Characterization of Visual Problems in Patients With Parkinson's Disease and Application of an Oculomotor and/or Perceptual Therapy Program"
Brief Title: " Visual Characterization of Parkinson's Patients and Oculomotor or Perceptual Therapy"
Status: Recruiting | Type: Observational
Sponsor: University of Valencia (Other)
Collaborators: Asociación Parkinson Valencia (Other); Hospital Arnau de Vilanova (Other)
Responsible Party: Principal Investigator, Amparo Diez, Principal Investigator, University of Valencia
Other Study IDs: 2161984
Record Dates: First submitted 2023-07-12; First posted 2023-09-11 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Vision; Ocular Motility Disorders; Perceptual Disorders
MeSH Terms: conditions — Parkinson Disease; Ocular Motility Disorders; Perceptual Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Parkinson Disease Group (PD): 1. Anamnesis
  2. Measurement of best visual acuity with an EDTRS (Early Treatment Diabetic Retinopathy Study) test
  3. Measurement of refraction with trial frame refraction
  4. Measurement of pupillary diameter under photopic and mesopic illumination conditions using a specific millimetric ruler
  5. Measurement of ocular sensory dominance with the red filter test
  6. Measurement of binocular vision status with the Cover Test, prism bar and Maddox wing
  7. Photopic and mesopic achromatic contrast sensitivity using the Functional Test Analyzer device
  8. Stereopsis using the Titmus Test
  9. Colour vision using the Farnsworth-Munsell 100 Hue sorting test
  10. Measurement of eye movements with aDEMd (adult Developmental Eye Movement) test and NSUCO (Northeastern State University College of Optometry)
  11. Measurement of reading speed with Radner-Vissum test
  12. National Eye Institute Visual Functioning Questionnaire-25 (NEI VFQ-25)
  Interventions: Other: Clinical measurements
- Control Group (GP): 1. Anamnesis: name, sex, date of birth, contact, family contact, medical report, Hoehn & Yahr classification, medication, systemic, ocular and family history, consumption of tobacco, alcohol, drugs, coffee, physical activity, eye colour, other observations
  2. Measurement of best visual acuity with an EDTRS test
  3. Measurement of refraction with trial frame refraction
  4. Measurement of pupillary diameter under photopic and mesopic illumination conditions using a specific millimetric ruler
  5. Measurement of ocular sensory dominance with the red filter test
  6. Measurement of binocular vision status with the Cover Test, prism bar and Maddox wing
  7. Photopic and mesopic achromatic contrast sensitivity using the Functional Test Analyzer device
  8. Stereopsis using the Titmus Test
  9. Colour vision using the Farnsworth-Munsell 100 Hue sorting test
  10. Measurement of eye movements with aDEMd test and NSUCO
  11. Measurement of reading speed with Radner-Vissum test
  12. NEI VFQ-25
  Interventions: Other: Clinical measurements
- Therapy Parkinson Disease Group (TPD): Oculomotor exercises such as tracking eye movements, saccadic eye movements and fixations will be performed. These exercises will be performed in a non-invasive manner using simple and easy-to-use instruments. An application on an electronic device, namely the virtual reality software Visionary, could also be used. If financial resources allow, the intention is to use tablets or computers for this purpose. Perceptual learning exercises will also be carried out on an electronic device. The following variables will be collected from these exercises: time taken to carry out the tests, errors made, speed of completion, latency, etc. These will be compared before and after the exercises in the third phase. In addition, the patients will be given indications for working on these exercises at home.
  Interventions: Other: Oculomotor or perceptual therapy
- Control Parkinson Disease Group (CPD): These patients will not receive oculomotor or perceptual therapy. They will be evaluated in the same manner as patients who will receive therapy, both at the beginning and at the end of therapy in the other group.
  Interventions: Other: Clinical measurements

INTERVENTIONS:
Other: Clinical measurements — Optometric measurements
  Groups: Control Group (GP); Control Parkinson Disease Group (CPD); Parkinson Disease Group (PD)
Other: Oculomotor or perceptual therapy — Oculomotor or perceptual visual learning exercices
  Groups: Therapy Parkinson Disease Group (TPD)

SUMMARY:
Parkinson's disease (PD) is the second most common neurodegenerative condition worldwide, characterised by motor symptoms, but with other symptoms such as visual impairment.

The aim is to compare visual function between PD patients and healthy subjects in order to adequately characterise the visual capabilities of the PD population and perform oculomotor or perceptual therapy to find optometric solutions to slow down the visual impairment they suffer from or minimise their visual symptoms.

In the first phase, non-invasive tests will be carried out, such as measuring visual acuity, refraction, pupil diameter in different lighting conditions, sensory dominance, contrast sensitivity, colour vision, stereopsis, reading speed, binocular vision, eye movements and influence on quality of life.

In the second, visual oculomotor or perceptual exercises will be performed in a group of PD patients to assess whether there is stabilisation of impairment or improvement of these visual skills. These will be performed in a non-invasive way using simple and easy-to-use instruments or an application on an electronic device could be used.

Finally, in the third phase, those visual skills that have been treated will be re-evaluated to assess possible changes, compared with a group of PD patients who have not undergone the visual exercises.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative condition worldwide. It is a movement disorder characterised by tremor, rigidity, bradykinesia and postural instability. However, 78% of PD patients report visual problems such as dry eye, reduced visual acuity, visual field defects, impaired contrast sensitivity (CS), impaired eye movements, diplopia, convergence insufficiency, impaired colour vision, visual hallucinations and problems in visual-spatial orientation. In fact, visual dysfunction is one of the initial symptoms of PD. A recent study has found that dopaminergic neurons affected in PD show physiological dysfunctions, but do not die. Currently, there is no cure for PD; treatments consist of controlling symptoms, and the earlier the disease is detected and administered, the more effective they are.

It is hypothesised that a programme of visual oculomotor therapy and/or visual perceptual learning (VPL) could slow or halt the deterioration of oculomotor ability and/or CS in these patients. Visual perceptual learning or VPL is a long-term improvement in performance on a visual task, any relatively permanent change in perception that arises from visual experience. Contrast Sensitivity or CS is the ability of the visual system to differentiate an object from the background in which it is located by the difference in contrast. It is the ability to detect differences in luminance between adjacent areas in an image.

If the results confirm the hypothesis, this study will have a great impact on the PD population because it could slow down the deterioration of oculomotor ability that 75% of them suffer from. It could also slow down the decline in CS that they suffer, as demonstrated by several studies. Consequently, patients would also experience an improvement in their quality of life, as they would be able to continue to perform activities of daily living that are affected by visual impairment such as walking, reading, driving and cooking. This would have a major impact on society as PD affects many people worldwide. In Europe, the prevalence and incidence rates of PD are estimated to be approximately 108-257/100 000 and 11-19/100 000 per year, respectively. Furthermore, this project would expand scientific knowledge because to date there is no literature that has evaluated VPL in patients with PD. However, there is research on amblyopia, Stargardt's disease and other neural pathologies, such as Huntington's disease. Likewise, with regard to oculomotor therapy, there is still a lot of research to be done, as there are few studies on this subject.

This is an analytical, longitudinal, prospective and observational study. In the first phase, to characterise the vision of the population with Parkinson's disease, non-invasive tests would be performed, such as measuring visual acuity, refraction, contrast sensitivity, colour vision, depth vision, the state of binocular vision and visual pathways and eye movements. Simultaneously, a control population will be measured to compare the data obtained in PD patients.

In a second phase, visual oculomotor and/or perceptual exercises would be performed in a group of PD patients to assess whether there is stabilisation of the impairment and/or improvement of these visual skills.

Finally, in the third phase, those visual skills that have been treated would be re-evaluated to assess possible changes, compared with a group of PD patients who have not undergone the visual exercises.

The research will be carried out at the Laboratory of Vision and Colour Sciences of the Department of Optics, Optometry and Vision Sciences of the University of Valencia, at the Arnau de Vilanova Hospital and at the Parkinson's Association of Valencia. These are the institutions from which the participants who take part in the study will come. They will do so voluntarily, will not be coerced to participate in any way and will be free to choose whether they want to participate or not, after having been explained to them what this project consists of. Furthermore, they will be able to revoke their signed consent at any time, so that they will automatically be excluded from the study and their data will not be used in the study if the patient so wishes. Furthermore, this project does not harm the patient's health and does not bring any financial benefit to the patient.

Only the members of the project will have access to the original study data. These data will be collected on paper, and the original source will be kept under lock and key in the laboratory of Vision and Colour Sciences of the Department of Optics, Optometry and Vision Sciences of the University of Valencia. For data analysis, the principal investigator will extract the data into a computer document in which each patient will be identified by a two-letter code (GP: control group; PD: Parkinson's patient) and three numbers. Not even the initials of the name will appear. Under this code, the data of each patient will be entered. This is the data that the rest of the group will see and have access to. Adverse event reporting and change management will be carried out through the Reservio platform, which will be used for appointment planning and online booking.

Data analysis will be carried out using the SPSS (Statistical Package for Social Sciences) statistical software and the Matlab numerical calculation system. The statistical analysis plan is as follows: the mean, standard deviation and normality of the samples will be performed with the Shapiro-Wilk test. Statistical comparison between groups will be performed with Student's t-test if the data follow a normal distribution or with the U-Mann-Whitney test otherwise. The statistical test used for qualitative variables will be Pearson's chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* Subjects without neurodegenerative diseases or systemic illnesses or ocular pathologies.
* Subjects not taking medication with visual side effects.
* Subjects able to perform the tests.
* Subjects of similar age and sex as their corresponding Parkinson's patient so that both samples are age and gender matched.
* Subjects diagnosed with Parkinson's disease.
* Parkinson's patients classified according to the Hoehn & Yahr Scale.

Exclusion Criteria:

* Subjects with ocular pathologies (such as Glaucoma, Age-Related Macular Degeneration, Retinopathies, Corneal Opacifications, Senile Cataracts, Severe Palpebral Ptosis) or systemic illnesses that may affect the visual system and alter the results (such as Severe Cardiopathies, Diabetes Mellitus, oncological diseases, systemic tissue disorders, chronic infectious diseases or conditions after organ or tissue transplantation).
* Subjects with neurodegenerative or neural diseases other than the study itself, such as Alzheimer's disease, Devic's disease, Huntington's disease, Creutzfeldt-Jakob disease, epilepsy, ataxia, multiple sclerosis or amyotrophic lateral sclerosis.
* Subjects taking medication that may alter any visual ability such as anxiolytics, antidepressants, sleeping pills.
* Subjects with problems in understanding and following the tests.
* Patients who have been previously treated under a vision therapy program.

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's Disease.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Anamnesis | 1 year
  Ocular and perceptual characterization of Parkinson's Disease visual capabilities with the following measurements (1-12).
  Anamnesis: Asking age, allergies, ocular and systemic pathologies, family background, current treatment (if proceed), consumption of tobacco, alcohol, drugs, coffee, tea, performance of physical activity, state on the Hoehn & Yahr classification, date of Parkinson's diagnosis and other observations.
Visual Acuity | 1 year
  Using an EDTRS (Early Treatment Diabetic Retinopathy Study) test for distance and near vision with the patient's optical correction, scale: LogMAR.
Refraction | 1 year
  Doing ocular compensation with trial frame refraction, units: diopters (D).
Pupillary diameter | 1 year
  Under photopic and mesopic illumination conditions using a specific millimetric ruler, units: millimeters (mm).
Ocular sensory dominance | 1 year
  Using the red filter test.
Binocular vision status | 1 year
  Using the Cover Test Cover Test, Modified Thorington Test Card to phoria measurement and fusional vergence measurement with prism bar, units: prismatic diopters (Δ).
Achromatic CSF (Contrast Sensitivity Funtion) | 1 year
  Under photopic and mesopic illumination conditions using the FACT (Funtional Acuity Contrast Test) test of the FVA (Functional Visual Analyzer) device of Stereo Optical Co., Inc.
Stereopsis | 1 year
  Using the Wirth points of the Titmus test, units: seconds of arc (").
Colour vision | 1 year
  Using the Farnsworth-Munsell 100 Hue sorting test and the Chromatic Threshold Measurement test.
Eye movements quality | 1 year
  Using aDEMd (adult Developmental Eye Movement with distractors) test and NSUCO (Northeastern State University College of Optometry) test. Units: seconds (s).
Reading speed | 1 year
  Using Radner-Vissum test, units: seconds (s).
Life quality assessment | 1 year
  Scoring the National Eye Institute Visual Functioning Questionnaire-25 (NEI VFQ-25). Higher scores mean a better outcome. Minimum value: 0, maximum value: 100.

SECONDARY OUTCOMES:
Pursuit eye movements | 1 year
  Would be performed noninvasively using simple, easy-to-use instruments such as flashlights, pointers, slates, Marsden's ball, rotating devices and Groffman's visual tracing test. If financial resources permit, an application on an electronic device could also be used.
  From these exercises, the following variables will be collected: time spent in the performance of the exercises in seconds (s) and errors made. These will be compared before and after the therapy.
  In addition, the patients would be given indications for the work of these exercises at home.
Saccadic eye movements | 1 year
  Would be performed noninvasively using simple, easy-to-use instruments such as flashlights, pointers, slates, Hart's charts, ARB charts and Ann Arbor tracing sheets. If financial resources permit, an application on an electronic device could also be used.
  From these exercises, the following variables will be collected: time spent in the performance of the exercises in seconds (s) and errors made. These will be compared before and after the therapy.
  In addition, the patients would be given indications for the work of these exercises at home.
Perceptual learning technique | 1 year
  Perceptual learning exercises could also be performed on an electronic device with a program that displays Gabor patches. This technique consists of a task with low-contrast, progressively decreasing, sustained attention, demanding and repetitive stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: María Amparo Díez-Ajenjo, PhD, Principal Investigator — University of Valencia
Locations (1):
- Hospital Arnau de Vilanova, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armstrong MJ, Okun MS. Diagnosis and Treatment of Parkinson Disease: A Review. JAMA. 2020 Feb 11;323(6):548-560. doi: 10.1001/jama.2019.22360. PMID 32044947
- [Background] Armstrong RA. Visual symptoms in Parkinson's disease. Parkinsons Dis. 2011;2011:908306. doi: 10.4061/2011/908306. Epub 2011 May 25. PMID 21687773
- [Background] Balestrino R, Schapira AHV. Parkinson disease. Eur J Neurol. 2020 Jan;27(1):27-42. doi: 10.1111/ene.14108. Epub 2019 Nov 27. PMID 31631455
- [Background] Beste C, Wascher E, Dinse HR, Saft C. Faster perceptual learning through excitotoxic neurodegeneration. Curr Biol. 2012 Oct 23;22(20):1914-7. doi: 10.1016/j.cub.2012.08.012. Epub 2012 Sep 13. PMID 22981772
- [Background] Borm CDJM, Visser F, Werkmann M, de Graaf D, Putz D, Seppi K, Poewe W, Vlaar AMM, Hoyng C, Bloem BR, Theelen T, de Vries NM. Seeing ophthalmologic problems in Parkinson disease: Results of a visual impairment questionnaire. Neurology. 2020 Apr 7;94(14):e1539-e1547. doi: 10.1212/WNL.0000000000009214. Epub 2020 Mar 11. PMID 32161030
- [Background] Campbell FW, Robson JG. Application of Fourier analysis to the visibility of gratings. J Physiol. 1968 Aug;197(3):551-66. doi: 10.1113/jphysiol.1968.sp008574. PMID 5666169
- [Background] Ekker MS, Janssen S, Seppi K, Poewe W, de Vries NM, Theelen T, Nonnekes J, Bloem BR. Ocular and visual disorders in Parkinson's disease: Common but frequently overlooked. Parkinsonism Relat Disord. 2017 Jul;40:1-10. doi: 10.1016/j.parkreldis.2017.02.014. Epub 2017 Feb 21. PMID 28284903
- [Background] Fahle M. Perceptual learning: a case for early selection. J Vis. 2004 Oct 26;4(10):879-90. doi: 10.1167/4.10.4. PMID 15595892
- [Background] Gonzalez-Rodriguez P, Zampese E, Stout KA, Guzman JN, Ilijic E, Yang B, Tkatch T, Stavarache MA, Wokosin DL, Gao L, Kaplitt MG, Lopez-Barneo J, Schumacker PT, Surmeier DJ. Disruption of mitochondrial complex I induces progressive parkinsonism. Nature. 2021 Nov;599(7886):650-656. doi: 10.1038/s41586-021-04059-0. Epub 2021 Nov 3. PMID 34732887
- [Background] Han G, Han J, Han K, Youn J, Chung TY, Lim DH. Visual Acuity and Development of Parkinson's Disease: A Nationwide Cohort Study. Mov Disord. 2020 Sep;35(9):1532-1541. doi: 10.1002/mds.28184. Epub 2020 Jul 25. PMID 32710579
- [Background] Huang CB, Zhou Y, Lu ZL. Broad bandwidth of perceptual learning in the visual system of adults with anisometropic amblyopia. Proc Natl Acad Sci U S A. 2008 Mar 11;105(10):4068-73. doi: 10.1073/pnas.0800824105. Epub 2008 Mar 3. PMID 18316716
- [Background] Kaur M, Saxena R, Singh D, Behari M, Sharma P, Menon V. Correlation Between Structural and Functional Retinal Changes in Parkinson Disease. J Neuroophthalmol. 2015 Sep;35(3):254-8. doi: 10.1097/WNO.0000000000000240. PMID 25807477
- [Background] Sasaki Y, Nanez JE, Watanabe T. Advances in visual perceptual learning and plasticity. Nat Rev Neurosci. 2010 Jan;11(1):53-60. doi: 10.1038/nrn2737. Epub 2009 Dec 2. PMID 19953104
- [Background] Sasso P, Silvestri V, Sulfaro M, Scupola A, Fasciani R, Amore F. Perceptual learning in patients with Stargardt disease. Can J Ophthalmol. 2019 Dec;54(6):708-716. doi: 10.1016/j.jcjo.2019.03.012. Epub 2019 May 31. PMID 31836104
- [Background] Savitt J, Aouchiche R. Management of Visual Dysfunction in Patients with Parkinson's Disease. J Parkinsons Dis. 2020;10(s1):S49-S56. doi: 10.3233/JPD-202103. PMID 32741840
- [Background] Shibasaki H, Tsuji S, Kuroiwa Y. Oculomotor abnormalities in Parkinson's disease. Arch Neurol. 1979 Jun;36(6):360-4. doi: 10.1001/archneur.1979.00500420070009. PMID 454234